CLINICAL TRIAL: NCT04442776
Title: Validation of a Dual Integrated Attention Program (DAIP) in People With Severe Dual Diagnosis Admitted to a Psychiatric Hospitalization Unit
Brief Title: Dual Integrated Attention Program (DAIP) in People With Severe Dual Diagnosis
Acronym: PAI-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Montse Cañabate, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Study DAIP; ESTUDIO PAI-D (Other: AEMPS(Agencia Española de Medicamentos))
Record Dates: First submitted 2020-02-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Diagnosis, Dual (Psychiatry)
Keywords: Psychiatric Dual Diagnosis; Integrated Attention; Program
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (Parallel Assignment)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will complete the Dual Integrated Attention Program (D-AIP) The D-AIP will consist on 6 individualized sessions with the psychiatric inpatients, and during follow-up up to one year after discharge in which 4 individual sessions and 3 telephone contacts will be made.
  Interventions: Behavioral: D-AIP
- Control group (No Intervention): The control group will complete the usual treatment. One session per day voluntary during admission and discharge, nursing consultations only to put injectable medication

INTERVENTIONS:
Behavioral: D-AIP — Intervention on change motivation, insight, medication adherence, drug consumption abstinence or reduction, therapeutic alliance, hopelessness and anxiety
  Arms: Intervention group

SUMMARY:
Aim: validate a Dual Integrated Attention Program (D-AIP) for mental health nursing in people with Severe Dual Diagnosis admitted to a psychiatric hospitalization unit

Design: Randomized Controlled Trial. Population: Inpatients with dual diagnosis.

DETAILED DESCRIPTION:
The main objective of the project is to validate a Dual Integrated Attention Program (D-AIP) for mental health nursing in people with Severe Dual Diagnosis admitted to a psychiatric hospitalization unit, assessing change motivation, insight, medication adherence, drug consumption abstinence or reduction, therapeutic alliance, hopelessness and anxiety, which this context generates. For this purpose, a randomized, prospective, one-year-longitudinal clinical trial will be conducted. This study will be applied on patients with diagnosis of schizophrenia, schizoaffective disorder and bipolar disorder types I and II who, after accepting to participate in the study and signing the informed consent, answer the PRISM questionnaire of admission in the hospitalization unit and fulfill the dual pathology criteria. After, they will be randomized in control group and intervention group (only the later will complete the D-AIP).

The D-AIP will consist on 6 individualized sessions with the psychiatric inpatients, and during follow-up up to one year after discharge in which 4 individual sessions and 3 telephone contacts will be made. In both groups, a different person from the one who performs the intervention and without knowledge of the group belonging will assess them with questionnaires in 9 moments during the whole follow-up year (Socrates 8D, Scale of Unawareness of Mental Disorder "SUMD", Morisky Medication Adherence Scale "MMAS-8", Working Alliance Inventory "WAI", Hamilton Anxiety Rating Scale "HARS" y Hopelessness Scale "HS") and will collect a urine sample in each evaluation. The sample size will be 86 subjects, for α=0.05 and power=0.80.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients diagnosed with some serious mental illness of the following:

   * Inpatients with diagnosis of schizophrenia
   * Inpatients with diagnosis schizoaffective disorder
   * Inpatients with diagnosis bipolar disorder types I
   * Inpatients with diagnosis bipolar disorder types II
2. Consumption of addictive substances

Exclusion Criteria:

* Intellectually Disabled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Stages of Change Readiness | 12 months
  Assessed by Questionnaire SOCRATES 8D
Insight | 12 months
  Assessed by Scale Unawareness of Mental Disorders (SUMD)
Medication Adherence | 12 months
  Assessed by Medication Adherence Scale (MMAS-8)
Therapeutic Alliance | 2-3 months
  Assessed by Working Alliance Inventory in patients and therapist (WAI-P and WAI-T)
Anxiety | 12 months
  Assessed by Hamilton Anxiety Rating Scale (HARS)
Hopelessness | 12 months
  Assessed by Hopelessness Scale (HS)

SECONDARY OUTCOMES:
Containments methods | 2-3 months
  Number of registered containments methods
Drug use change | 12 months
  Presence of drug abuse through a urine sample with "10-panel drug test"
Hospital readmissions | 12 months
  Number of registered hospital readmissions
Dual diagnosis knowledge | 12 months
  Assessed by ad-hoc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Montse Cañabate, Dra., Principal Investigator — Cardenal Herrera University